CLINICAL TRIAL: NCT04122313
Title: Efficacy of Post-contracture Release Radiation for the Treatment of Dupuytren's Disease
Brief Title: Post-contracture Release Radiation for Dupuytren's Disease
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ORTHOSURG-2018-26681
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Dupuytren's Disease; Dupuytren Contracture; Dupuytren Disease of Palm and Finger; Dupuytren Disease of Finger; Dupuytrens Contracture of Both Hands; Dupuytren's Disease of Palm of Right Hand; Dupuytren's Disease of Palm of Left Hand; Dupuytren Contracture of Right Palm; Dupuytren Contracture of Left Palm; Dupuytren's Contracture Left; Dupuytren's Contracture Right
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Dupuytren's Contracture Disease: Patients with Dupuytren's Disease following the current treatment pathway
  Interventions: Other: Evaluation of Dupuytren's Disease Treatment

INTERVENTIONS:
Other: Evaluation of Dupuytren's Disease Treatment — There are no study interventions. The study interaction will be asking the patients to complete an additional outcome questionnaire and allow a medical record review.

SUMMARY:
To determine if the clinical impression of clinicians, ie that patients are improving with the current treatment pathway for Dupuytren's (contracture release followed by radiation), can be substantiated with scientific evidence.

DETAILED DESCRIPTION:
This is an observational, pilot study. Participants will be treated according to a standard treatment pathway, which includes contracture release treatment modalities such as limited fasciectomy, PNA and CCH injection, followed by post-operative radiation. All enrolled participants will undergo radiation treatment as soon as possible following contracture release. Radiotherapy will consist of 5 daily treatments of 300 cGy delivered to the palmar area followed by a 6-8 weeks break then a second 5 day course of radiation at 300 cGy, for a total of 3000 cGy in 10 total fractions. This dosing schedule is commonly used in the published literature. The data to be collected about participants, is their Southampton Dupuytren's score, history and clinical symptoms and photographs of their hand. This information will be obtained at baseline (pre-surgical intervention), at radiation treatment planning, approximately 6 weeks after completion of all radiation and at 1 and 2 years following completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of Dupuytren's disease
* English-speaking

Exclusion Criteria:

- Patients with Dupuytren's disease who are not currently seeking treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English-speaking adults with a diagnosis of Dupuytren's disease whose have chosen to follow the current treatment pathway.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Southampton Dupuytren's Scoring System (SDSS) Questionnaire | 2 years
  The primary study endpoint is the patient's self-reported function which will be assessed using the validated Southampton Dupuytren's Scoring System (SDSS) questionnaire. The SDSS is a 5 item questionnaire with item scores ranging from 0 (no problem) to 4 (severe problem). Total scores are a sum of the 5 item scores with a total score range of 0 to 20. High scores indicate greater impairment due to the disease.

SECONDARY OUTCOMES:
Common Terminology Criteria for Adverse Events (CTCAE) | 2 years
  The secondary endpoint will be the recurrence rate (which is defined as an increase in joint contracture on any treated joint of at least 20 degrees at one year post-treatment compared to six weeks post treatment) and skin toxicity, which will be assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Chang, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No